CLINICAL TRIAL: NCT01371253
Title: 10 Weeks of NIntendo wIi Fit balanCe Training Improved Postural balANce and Muscle Strength in Elderly Individuals: Double Blinded, Randomised Controlled Trial
Brief Title: 10 Weeks of NIntendo wIi Fit balanCe Training Improved Postural balANce and Muscle Strength in Elderly Individuals
Acronym: WIICAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Martin Joergensen, Cand. scient.,Ph.d. Student, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Wii1
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Impaired Balance
Keywords: Nintendo wii; postural balance; muscle strength; elderly

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nintendo Wii traning (Experimental): Balance training
  Interventions: Other: Nintendo wii balance training
- EVA-soles (Placebo Comparator)
  Interventions: Other: EVA-soles

INTERVENTIONS:
Other: Nintendo wii balance training
  Arms: Nintendo Wii traning
Other: EVA-soles
  Arms: EVA-soles

SUMMARY:
On a yearly basis roughly 40.000 individuals aged 65+ contact the emergency departments in Denmark as a result of an accidental fall, and in about 30% of these cases hospitalization is required. The cost of these admissions vary according to the type of injury with hip fractures being the most expensive accident {{113 Chrischilles,E. 1994; }}. The total average cost of a severe hip fracture in the Danish healthcare system resulting in nursing home placement has been estimated to approximately 365.000 Danish Kroner (Dkk) per year {{288 Christensen,P.M. 2005;}}. In addition, about 20 % of the elderly individuals who sustain a hip fracture will die within 6 months {{200 Brot,C. 2006; }}. For the society the outcome of falling in the elderly population is therefore not only associated with severe human but also economical consequences. Hence, it is essential to refine, develop and think "out of the box" when future intervention programs are designed and employed in the elderly community.

One such "out of the box" intervention could be balance training with a Nintendo Wii Fit board (Nintendo Wii, Nintendo Co Ltd, Minami-ku Kyoto, Japan). The Nintendo Wii Fit board is a new generation of computer game which uses 3D tracking of the participants' motion and gestures. This means that the user interacts in and controls elements of the 3D gaming world with their own body {{307 LaViola,J.J.,Jr 2008;}}. In the case of the Wii Fit board, it detects the body sway and center of pressure (COP) of the participant and displays it onto a TV screen in different balance sceneries. A virtual character on the TV then reacts according to the user's movement and gesture (ex. skiing down a ski slope passing thru gates). This enables the user to perform tasks that, they may not be able to execute safely or at all in real-world situations. Interestingly in this context a study by Sihvonen et al from 2004 showed a compliance of 97,5% using the same technique as the Wii Fit only in 2D and with a poor graphical display. Further, the Sihvonen-study showed that 2D "biofeedback" intervention of only 4 weeks proved successful in terms of improved postural balance, physical activity and life quality {{297 Sihvonen,S. 2004;}}. Finally, traditional methods when promoting physical activity in the elderly population has been limited by lack of motivation or poor compliance (REFS), which possibly has prevented the elderly from reaching a maximum rehabilitation potential(REFS). Furthermore, in the follow-up period after these traditional intervention studies, it has been documented how difficult it is for the elderly to sustain the same training volume on themselves (REFS).

Virtual reality systems like the Nintendo Wii Fit have been developed specifically for rehabilitation of the upper- {{301 Kuttuva,M. 2006;300 Dvorkin,A.Y. 2006;}} and lower-extremities and gait training {{298 Deutsch,J.E. 2007;}}. Further virtual reality platforms have been use for rehabilitation and training of reaching movements {{302 Piron,L. 2001;}}, motor coordination {{303 Broeren,J. 2002;}}, hand strength and range of motion, speed of hand movement{{304 Jack,D. 2001;305 Merians,A.S. 2002;}}. But so far most of these systems have not become commercially available possible due to a very high cost {{294 Deutsch,J.E. 2008;}}. Moreover in some cases the virtual rehabilitation environment has to be constructed from scratch making the hole process and implication very complicated {{306 Weiss,P.L. 2004;}}. Thus, designing an intervention program that utilizes the low-cost ready-to-use Wii Fit platform could be a possible research direction to explore. At the moment few studies have been conducted using the Nintendo Wii console. Among the few some have investigated the energy expenditure in kids (11-17 years of age) playing Wii Sports (bowling, tennis and boxing) compared to sedentary xbox games and actual bowling, tennis and boxing {{ 295 Graves,L.E. 2008; 296 Graves,L. 2008; }} while others have explored the Nintendo Wii console for rehabilitation of an adolescent with cerebral palsy {{294 Deutsch,J.E. 2008; }}.

To the authors knowledge no studies have investigated the effect of 10 weeks of Nintendo Wii Fit balance training in seniors (+65 years). The main purpose of the study is to investigate the hypothesis: That 10 weeks of Nintendo Wii Fit balance training in a group of seniors (+65 years of age) have a significant effect on postural balance and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Age above 65 years
* No physical therapy during the previous month
* capable of understanding instructions
* not recovering from acute illness
* minimal loss of visual acuity
* Selfprecived balance (good, average, poor) = average or poor
* No orthopaedic Surgery within the last 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Balance | Baseline=june; Endline=september
  M-L sway velocity, A-P sway velocity and velocity moment on a Metitur, FI " Good Balance"
Muscle strength | Baseline=june; Endline=september
  Maximum muscle strength (MVC) and rate of force development (RFD) bilateral assessed on a Newtest,FI legpress
Motivation | Baseline=june; Endline=september
  At the end of the study 3 questions on the likert scale will be asked in order to evaluate the participants motivation for further nintendo wii training.

SECONDARY OUTCOMES:
Fear of falling | Baseline=june; Endline=september
  Fear of falling will be assessed using the FES-I (short)
Timed up and go | Baseline=june; Endline=september
  The TUG test

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg Hospital, Aalborg, North Denmark, Denmark

REFERENCES:
- [Derived] Jorgensen MG, Laessoe U, Hendriksen C, Nielsen OB, Aagaard P. Efficacy of Nintendo Wii training on mechanical leg muscle function and postural balance in community-dwelling older adults: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2013 Jul;68(7):845-52. doi: 10.1093/gerona/gls222. Epub 2012 Oct 31. PMID 23114461